CLINICAL TRIAL: NCT06963840
Title: Effect of Theronomic Ova-All Care on Biomarkers of Ovarian Health in Adult Female With Polycystic Ovarian Syndrome
Acronym: Ova-All Care
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wellizen Australia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WEL202501
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Polycystic Ovarian Syndrome (PCOS)
Keywords: probiotic; prebiotic; postbiotic; ovary; menstruation; polycystic ovarian syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Theronomic Ova-All Care (Experimental): Active treatment - Theronomic Ova-All Care
  Interventions: Dietary Supplement: Theronomic Ova-All Care

INTERVENTIONS:
Dietary Supplement: Theronomic Ova-All Care — Two capsules of Theronomic Ova-All Care, one a day, for 12 weeks. Ova-All Care is a tribiotic, a health product that includes prebiotics, probiotics, and postbiotics. Ova-All Care affects ovarian health by regulating the gut microbiome, which affects oestrogen production and other factors.

SUMMARY:
Theronomic Ova-All Care is a tribiotic health product aimed at improving ovarian health in people with polycystic ovarian syndrome (PCOS). In this study, a total of 16 participants with PCOS diagnosed by a gynaecologist will be invited to take Ova-All Care, two capsule once a day, for 12 weeks. Biomarkers of ovarian health will be measured at baseline, four weeks after the start of the intervention, and at the end of the intervention.

ELIGIBILITY:
Inclusion criteria

1. Women aged 18-40 years
2. Previous diagnosis of PCOS by a gynaecologist
3. Able to take body temperature every day for 12 weeks
4. Able to attend the testing centre every 4 weeks
5. Able to complete online questionnaires

Exclusion criteria

1. Pregnancy, lactation;
2. Uterine amenorrhea (such as intrauterine adhesions)
3. Thyroid disease or hyperprolactinemia
4. Liver and kidney dysfunction, autoimmune diseases (such as systemic lupus erythematosus), malignant tumors, mental illness
5. Use of contraceptives, hormone replacement therapy (HRT), immunosuppressants and other drugs that affect ovarian function in the past 3 months.
6. Smokers (>5 cigarettes per day), alcoholics;
7. Unable to cooperate with follow-up or refuse to sign informed consent.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-05-09 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Serum oestrogen level | From enrollment to end-of intervention (Week 12)
  Serum oestrogen levels determined by blood test, pg/mL
  We will conduct two subgroup analyses with participants with excessively low (less than 25 pg/mL) and excessively high (more than 138 pg/mL) serum oestrogen levels

SECONDARY OUTCOMES:
HbA1c | From enrollment to end-of intervention (Week 12)
  Haemoglobin A1c in percentage.
  We will conduct a subgroup analysis with participants who have an abnormal HbA1c (more than 5.9%) at baseline.
Fasting Blood Glucose | From enrollment to end-of intervention (Week 12)
  Fasting Blood Glucose (FBG), in mmol/L
  We will conduct a subgroup analysis with participants who have an abnormal FBG (more than 6.22 mmol/L) at baseline.
Insulin | From enrollment to end-of intervention (Week 12)
  Serum insulin level, μU/mL.
  We will conduct a subgroup analysis with participants who have an abnormal insulin (more than 24.8 μU/mL) at baseline.
HOMA-IR | From enrollment to end-of intervention (Week 12)
  Homeostatic Model Assessment of Insulin Resistance, no unit.
  We will conduct a subgroup analysis with participants who had abnormal HOMA-IR (more than 2.0) at baseline.
LH | From enrollment to end-of intervention (Week 12)
  Luteinising hormone, in IU/L.
  We will conduct a subgroup analysis with participants who had abnormal LH (more than 11.6) at baseline.
LH/FSH | From enrollment to end-of intervention (Week 12)
  Ratio of luteinising hormone on follicle-stimulating hormone.
  We will conduct a subgroup analysis with participants who had abnormal LH/FSH (more than 2.0) at baseline.
Progesterone | From enrollment to end-of intervention (Week 12)
  Progesterone level, ng/mL.
  We will conduct a subgroup analysis with participants who had abnormal progesterone (more than 2.1) at baseline.
Testosterone | From enrollment to end-of intervention (Week 12)
  Testosterone levels, ng/mL
  We will conduct a subgroup analysis with participants who had abnormal testosterone (more than 0.55 ng/mL) at baseline.
Weight | From enrollment to end-of intervention (Week 12)
  Weight measured by a weight scale, in kg
  We will conduct two subgroup analyses with participants who are overweight (more than 25 kg/m2) and obese (more than 30 kg/m2) at baseline, respectively.
BMI | From enrollment to end-of intervention (Week 12)
  Body Mass Index, calculated based on the weight and height, in kg/m2.
  We will conduct two subgroup analyses with participants who are overweight (more than 25 kg/m2) and obese (more than 30 kg/m2) at baseline, respectively.
Waist size | From enrollment to end-of intervention (Week 12)
  Waist size measured with a measuring scale, in cm.
  We will conduct a subgroup analyses with participants who had an excessive waist circumference (more than 80 cm) at baseline.
Buttocks size | From enrollment to end-of intervention (Week 12)
  Buttocks size measured with a measuring scale, in cm.
  We will conduct a subgroup analyses with participants who had an excessive buttocks circumference (more than 93 cm) at baseline.
Thigh size | From enrollment to end-of intervention (Week 12)
  Thigh size measured with a measuring scale, in cm.
SBP | From enrollment to end-of intervention (Week 12)
  Systolic blood pressure, in mmHg.
  We will conduct a subgroup analyses with participants who had an excessive SBP (more than 120 mmHg) at baseline.
DBP | From enrollment to end-of intervention (Week 12)
  Diastolic blood pressure, in mmHg.
  We will conduct a subgroup analyses with participants who had an excessive DBP (more than 90 mmHg) at baseline.
Total Cholesterol | From enrollment to end-of intervention (Week 12)
  Total cholesterol, in mmol/L.
  We will conduct a subgroup analyses with participants who had an excessive total cholesterol (more than 5.6 mmol/L) at baseline.
Triglycerides | From enrollment to end-of intervention (Week 12)
  Triglycerides, in mmol/L.
  We will conduct a subgroup analyses with participants who had excessive triglycerides (more than 2.3 mmol/L) at baseline.
LDL | From enrollment to end-of intervention (Week 12)
  Low density lipoprotein, in mmol/L.
  We will conduct a subgroup analyses with participants who had an excessive waist circumference (more than 4.11 mmol/L) at baseline.
HDL | From enrollment to end-of intervention (Week 12)
  High density lipoprotein, in mmol/L.
  We will conduct a subgroup analyses with participants who had an excessive HDL (less than 1.15 mmol/L) at baseline.
hsCRP | From enrollment to end-of intervention (Week 12)
  high-specificity C-reactive protein, in mg/L.
  We will conduct a subgroup analyses with participants who had an excessive hsCRP (more than 4 mg/L) at baseline.
Rotterdam criteria on ultrasound | From enrollment to end-of intervention (Week 12)
  Yes/No, must meet at least of the of following criteria on one ovary for "Yes"
  1. ≥20 follicles per ovary, measuring 2-9 mm in diameter,
     OR
  2. Ovarian volume >10 mL
Cyst number | From enrollment to end-of intervention (Week 12)
  Number of cysts measured by ultrasound, in numbers
Cyst size | From enrollment to end-of intervention (Week 12)
  Size of the largest cyst, measured by ultrasound, in mm
Endometrial thickness | From enrollment to end-of intervention (Week 12)
  Endometrial thickness, measured with ultrasound, in mm
Normal ultrasound | From enrollment to end-of intervention (Week 12)
  Normal/abnormal ultrasound, based on the ultrasound report, dichotomous data
Menstrual cycle length | From enrollment to end-of intervention (Week 12)
  length of the menstrual cycle, assessed with a tracking app, in days
Normal menstrual cycle | From enrollment to end-of intervention (Week 12)
  Dichotomous data Normal = 21-35 Abnormal: more than 35 days or less than 21 days
Menstruation duration | From enrollment to end-of intervention (Week 12)
  Menstruation assessed with a self-reported questionnaire, in days
Menstrual pain | From enrollment to end-of intervention (Week 12)
  Average level of menstrual pain on a scale of 0 to 10, 10 being the most severe possible pain. No unit.
Maximal menstrual pain | From enrollment to end-of intervention (Week 12)
  Maximal level of pain experienced during menstruation, assessed with a participant-reported questionnaire, on a scale of 0 to 10, 10 being the most severe possible pain. No unit.
Quantity of menstruation | From enrollment to end-of intervention (Week 12)
  Quantity of blood in the menstruation, assessed with a participant-reported questionnaire, on a Lickert scale with 5 options: too scarce, relatively scarce, normal, relatively abundant and too abundant. In points (0 to 4).
Ovulation during last cycle | From enrollment to end-of intervention (Week 12)
  Dichotomous Ovulation: A significant increase in BBT of around 0.3°C to 0.6°C observed between the follicular and luteal phases.
  No ovulation: no bi-phasic feature.
Left ovary volume | From enrollment to end-of intervention (Week 12)
  Left ovary volume in mL.
  We will conduct a subgroup analysis with participants who had an abnormal left ovary size (more than 10 mL) at baseline.
Right ovary volume | From enrollment to end-of intervention (Week 12)
  Right ovary volume in mL.
  We will conduct a subgroup analysis with participants who had an abnormal right ovary size (more than 10 mL) at baseline.
Ovulation | Baseline to end-of-intervention
  Number of participants who ovulated during their last cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Pony Testing Centre, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
We will consider sharing IPD upon reasonable request